CLINICAL TRIAL: NCT04170491
Title: The Use of Continuous Electroencephalographic (EEG) Monitoring for Cases of Refractory Status Epilepticus: Does it Affect the Final Patient Outcome
Brief Title: EEG Monitoring for Refractory Status Epilepticus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 240176
Record Dates: First submitted 2019-11-01; First posted 2019-11-20 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Status Epilepticus
MeSH Terms: conditions — Status Epilepticus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): The standard medical care (Control) group will receive sequential portable EEGs, performed according to clinical demand. These patients usually have 2 recordings of 20-30 minutes each within 24 or 48 hours. The studies include baseline recoding and recording after auditory, tactile and nociceptive stimulation. The EEGs will be visually reviewed and reported within 4 hours after the recording completion by a Consultant Clinical Neurophysiologist or other doctor with equivalent qualifications.
- cEEG (Experimental): The treatment (cEEG) group will have cEEG applied within 12 hours of RSE diagnosis, which will continue until 24 hours after cessation of clinical and electrical seizure activity. Reactivity testing with auditory, tactile and nociceptive stimulation will be repeated at least once daily. The cEEG will be visually interpreted twice daily by a Consultant Clinical Neurophysiologist and the results will be communicated within two hours of their completion to the treating clinical team.
  Interventions: Diagnostic Test: Continuous EEG

INTERVENTIONS:
Diagnostic Test: Continuous EEG — Continuous EEGs will be performed with 21 electrodes and polygraphy (ECG and EMG) placed according to the international 10-20 system. In case of extensive neurosurgical defects, a reduced montage may be applied in patients from either group. This information will be added in CRF. The reduced montage in these cases is not expected to reduce the diagnostic accuracy and the outcome, as the neurophysiological changes are generally diffuse and will be detected by adjacent electrodes.
  Arms: cEEG

SUMMARY:
This is a prospective randomized study to investigate the yield of continuous electroencephalogram (cEEG), as a diagnostic tool in intensive care unit (ICU), for patients with refractory status epilepticus (RSE) and the contribution of this test to the patient final outcome, compared with standard medical care. Specifically, the hypothesis is that the use of cEEG for patients with RSE will significantly reduce the length of in-hospital stay, mortality, and subsequent complications (such as infections or pressure ulcers). It is also predicted that quality of life will be higher following cEEG at 0, 3, 6 and 12 months after discharge. As there are currently no data available from previous studies assessing the impact of cEEG on markers of the final clinical outcome in patients with RSE, this study is going to start as a feasibility study, aiming to obtain initial data for the primary outcome measure, in order to perform a sample size calculation for a larger future trial. The pilot study will also assess the integrity of the study protocol, specifically the recruitment process and the consent procedure, and also determine the necessary costs for running a cEEG service in ICU for patients with RSE

DETAILED DESCRIPTION:
The study is a randomised feasibility study.

The patients participating in the study will be randomised 1:1 in two groups. The randomisation will be stratified by three status epilepticus (SE) aetiologies a) previous epilepsy b) acute central nervous system insult c) cryptogenic/ unknown.

The standard medical care group (Control group) will receive sequential portable electroencephalograms (EEGs), performed according to the clinical demand. The treatment group (cEEG group) will have cEEG, which will continue until 24 hours after cessation of clinical and electrical seizure activity. The patients will be treated by the same medical team of neurologists or neurointensivists, according to the same guidelines.

Clinical data will be collected from observation of in-patient medical records. The information will include demographics i.e. age, gender and ethnicity group, information about previous medical history and specifically previous history of epilepsy. The investigators will record the type of epilepsy, the type of previous seizures, their frequency, previous admissions due to SE and current and previously used antiepileptic drugs. These data can be obtained either by the patient or the next of kin and if the patient is followed up in the local epilepsy service, the required data may be obtained from the medical records.

Regarding the acute presentation of status epilepticus, data will be collected regarding the date and the time of diagnosis of SE, the date of seizure onset, the level of consciousness on presentation, the type of seizures during SE (i.e. focal motor, generalised motor, absence etc) and SE aetiology, if available. If the SE is diagnosed by EEG as non-convulsive, the date of the diagnosis will be recorded. The types of seizures during the course of SE will be recorded, as well as the antiepileptic drugs and sedation used, including the doses. The SE severity score (STESS) will be calculated early during the patient admission to ICU. The date that the patient was fit for discharge from ICU will be obtained, as well as the date of discharge from hospital. It is noted that the date the patient is fit for discharge from ICU is not always the same as the actual date of ICU discharge. The data will also include in-hospital and 30-days mortality, the time until seizure control and the reported hospital acquired complications and specifically healthcare-associated infections, pressure injuries, falls resulting in fractures or injuries, respiratory complications, venous thromboembolism and medication complications. The quality of life index will be assessed with the health questionnaire introduced by EuroQol Group (version EQ-5D-5L), at 0, 3 ,6 and 12 months post discharge and/ or the Quality of Life in Epilepsy questionnaire (QOLIE), which will be mailed to the patients. If the patient is not able to provide this information in writing, these data will be collected with brief telephone interview.

The observational data will be collected by the research nurse and will be transferred to the case report form (CRF). The specific information, regarding the seizure types and the seizure aetiology, will require input from the medical team and specifically the neurologist, the neurointensivist and the clinical neurophysiologist. The information gather will be reviewed and supervised by the Principal Investigator (PI).

The data regarding the hospital costs for each patient will be collected after the patient's discharge and will be based on the specific coding of all medical, diagnostic and therapeutic interventions registered for each patient, taking into account the additional time required for assessing cEEG data. The clinical neurophysiologist and the physiologist will log their clinical activity time required for reviewing the cEEG recordings.

The data will be transferred to CRF and the length of ICU and in-hospital stay and the quality of life measures will be compared between groups in order to identify differences in the final outcome between the control and the cEEG groups. Similarly, the costs for management of the two patient groups will be compared.

The calculation of the sample size for the larger study will be performed after the collection of 40 cases.

ELIGIBILITY:
Inclusion Criteria:

* • Patients aged > 16 years

  * Consent obtained according to Mental Capacity Act 2005
  * Patients admitted to ICU for treatment of status epilepticus or admitted for another reason and diagnosed with SE during their admission
  * Convulsive Status epilepticus defined by either:

    * Tonic-clonic SE lasting longer than 5 minutes,
    * Focal SE with impaired consciousness lasting longer than 10 minutes
    * or Non-Convulsive SE according to Salzburg consensus criteria
  * Status epilepticus that continues despite treatment with benzodiazepine and one antiepileptic medication

Exclusion Criteria:

* Anoxic brain injury

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-03-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Length of ICU stay | 18 months from recruitment onset (anticipated)
  The length of ICU stay will be measured as the primary outcome measure. This will be compared between the two groups.

SECONDARY OUTCOMES:
Health status evaluation | End of the study- 3 years
  Assessed with EQ-5D-5L scale. Maximum value 1 indicates reported full health state. Minimum value -0.594.
Mortality | 18 months from recruitment onset
  In-hospital and/or 30-days mortality
Hospital charges | End of the study- 3 years
  The hospital charges (in British pounds) will be compared between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No